CLINICAL TRIAL: NCT02083679
Title: A Phase Ib, Open-label, Dose Escalation Trial Investigating Different Doses and Schedules of Sym004 in Combination With Platinum-doublets in Subjects With Stage IV Non-small Cell Lung Cancer
Brief Title: Sym004 in Subjects With Stage IV Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor the return rights of the compound to the collaboration partner for further clinical development
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR200637-003; 2013-003995-11 (EudraCT Number)
Record Dates: First submitted 2014-03-07; First posted 2014-03-11 (Estimated); Results first posted 2016-10-25 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Carcinoma, Non-Small-Cell Lung; Sym004
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Gemcitabine; Pemetrexed; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Part 1: Sym004 6 mg/kg + Cisplatin/Gemcitabine (Experimental)
  Interventions: Drug: Part 1: Sym004 6 mg/kg + Cisplatin/Gemcitabine
- Part 1: Sym004 6 mg/kg + Cisplatin/Pemetrexed (Experimental)
  Interventions: Drug: Part 1: Sym004 6 mg/kg + Cisplatin/Pemetrexed
- Part 1: Sym004 6 mg/kg + Carboplatin/Paclitaxel (Experimental)
  Interventions: Drug: Part 1: Sym004 6 mg/kg + Carboplatin/Paclitaxel
- Part 1: Sym004 6/12 mg/kg + Carboplatin/Paclitaxel (Experimental)
  Interventions: Drug: Part 1: Sym004 6/12 mg/kg + Carboplatin/Paclitaxel

INTERVENTIONS:
Drug: Part 1: Sym004 6 mg/kg + Cisplatin/Gemcitabine — Sym004 will be administered as an intravenous infusion at a dose of 6 mg/kg weekly until unacceptable toxicity, progressive disease, withdrawal of consent, or until the subject meets any of the criteria for subject withdrawal, or withdrawal from the investigational medicinal product (IMP) in combination with platinum-doublet chemotherapy regimen of cisplatin/gemcitabine (cisplatin 75 mg/m^2 on Day 1 plus gemcitabine 1250 mg/m^2 on Days 1 and 8 of every 3-Week cycle intravenously for a maximum of 6 treatment cycles).
  Arms: Part 1: Sym004 6 mg/kg + Cisplatin/Gemcitabine
Drug: Part 1: Sym004 6 mg/kg + Cisplatin/Pemetrexed — Sym004 will be administered as an intravenous infusion at a dose 6 mg/kg weekly until unacceptable toxicity, progressive disease, withdrawal of consent, or until the subject meets any of the criteria for subject withdrawal, or withdrawal from the IMP in combination with platinum-doublet chemotherapy regimen of cisplatin/pemetrexed (cisplatin 75 mg/m^2 plus pemetrexed 500 mg/m^2 on Day 1 of every 3-Week cycle intravenously for a maximum of 6 treatment cycles).
  Arms: Part 1: Sym004 6 mg/kg + Cisplatin/Pemetrexed
Drug: Part 1: Sym004 6 mg/kg + Carboplatin/Paclitaxel — Sym004 will be administered as an intravenous infusion at a dose 6 mg/kg weekly until unacceptable toxicity, progressive disease, withdrawal of consent, or until the subject meets any of the criteria for subject withdrawal, or withdrawal from the IMP in combination with platinum-doublet chemotherapy regimen of carboplatin/paclitaxel (carboplatin area under the concentration-time curve (AUC) = 6 milligram per millilitre per minute [mg/mL/min] plus paclitaxel 225 mg/m^2 on Day 1 of 3-Week cycle intravenously for a maximum of 6 treatment cycles).
  Arms: Part 1: Sym004 6 mg/kg + Carboplatin/Paclitaxel
Drug: Part 1: Sym004 6/12 mg/kg + Carboplatin/Paclitaxel — Sym004 will be administered as an intravenous infusion at a dose 6 mg/kg on Day 1 and 12 mg/kg on Day 8 of a 3-Week cycle until unacceptable toxicity, progressive disease, withdrawal of consent, or until the subject meets any of the criteria for subject withdrawal, or withdrawal from the IMP in combination with platinum-doublet chemotherapy regimen of carboplatin/paclitaxel (carboplatin AUC = 6 mg/mL/min plus paclitaxel 225 mg/m^2 on Day 1 of every 3-Week cycle intravenously for a maximum of 6 treatment cycles).
  Arms: Part 1: Sym004 6/12 mg/kg + Carboplatin/Paclitaxel

SUMMARY:
This is a multi-center, open-label, Phase 1b, dose escalation trial of Sym004 administered in combination with 1 of 3 platinum-doublets in subjects with Stage IV Non-Small Cell Lung Cancer (NSCLC).

The sponsor decided to discontinue the development of Sym004. Also the decision was made to discontinue the development of Sym004 in NSCLC indication. The decision to discontinue Sym004 in NSCLC was not related to any safety or efficacy findings regarding Sym004. As a result of the early discontinuation of the trial during the dose escalation part, the expansion cohort will no longer be performed hence the pre-specified secondary endpoints are not analyzed and were removed from the protocol based on protocol amendment 2 dated 31 March 2015.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients (except where inpatient stay is required for medical need at the Investigator's discretion) at least 18 years of age at the time of informed consent
* Histologically-confirmed NSCLC Stage IV disease (according to the seventh edition of the lung cancer staging system)
* Eligibility for platinum-based chemotherapy
* Tumor tissue available for epidermal growth factor receptor (EGFR) expression analysis
* Measurable disease defined as 1 or more target lesions according to Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST 1.1)
* Life expectancy of at least 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 1
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Previous therapy for Stage IV NSCLC, or neo- or adjuvant chemotherapy or chemoradiotherapy within the previous 6 months
* Previous investigational drug or any anticancer therapy in the 30 days (or 5 half-lives for non-cytotoxics, whichever is shorter) prior to the start of trial treatment
* In countries where anaplastic lymphoma kinase (ALK) inhibitors are available for the treatment of NSCLC, subjects need to have been screened for ALK fusion gene rearrangements and excluded if positive, unless previously treated and progressed on an appropriate tyrosine kinase inhibitor (TKI) therapy
* In countries where EGFR TKIs are available for the treatment of NSCLC, subjects need to have been screened for EGFR mutations and excluded if positive, unless previously treated and progressed on an appropriate TKI therapy
* Concurrent chronic immunosuppressive or hormone anticancer therapy (except other physiologic hormone replacement)
* Known brain metastases (unless asymptomatic and treated) or leptomeningeal metastases, including suspected leptomeningeal spread with positive cytology
* History of any other malignancy within 5 years (except basal cell carcinoma of the skin or carcinoma in situ of the cervix)
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (2):
- Please Contact U.S. Medical Information Located in, Rockland, Massachusetts, United States
- Please contact the Merck KGaA Communication Center located in, Darmstadt, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 5 clinical trial sites within France and the United States. First subject first visit: 03 July 2014 and last subject last visit: 31 August 2015. Clinical data cut-off date: 16 September 2015
Pre-assignment Details: This study was planned to be conducted in 2 parts; Part 1 was the dose escalation part and Part 2 was the expansion cohort. However, due to premature termination of the trial by the Sponsor, the Expansion Cohort (Part 2) was not conducted.
Groups:
- Part 1: Sym004 6 mg/kg + Cisplatin/Gemcitabine: Sym004 administered as an intravenous infusion at a dose of 6 milligram per kilogram (mg/kg) weekly until unacceptable toxicity, progressive disease, withdrawal of consent, or until the subject met any of the criteria for subject withdrawal, or withdrawal from the investigational medicinal product (IMP) in combination with platinum-doublet chemotherapy regimen of cisplatin/gemcitabine (cisplatin 75 milligram per meter square (mg/m^2) on Day 1 plus gemcitabine 1250 mg/m^2 on Days 1 and 8 of every 3-Week cycle intravenously for a maximum of 6 treatment cycles).
- Part 1: Sym004 6 mg/kg + Cisplatin/Pemetrexed: Sym004 administered as an intravenous infusion at a dose 6 mg/kg weekly until unacceptable toxicity, progressive disease, withdrawal of consent, or until the subject met any of the criteria for subject withdrawal, or withdrawal from the IMP in combination with platinum-doublet chemotherapy regimen of cisplatin/pemetrexed (cisplatin 75 mg/m^2 plus pemetrexed 500 mg/m^2 on Day 1 of every 3-Week cycle intravenously for a maximum of 6 treatment cycles).
- Part 1: Sym004 6 mg/kg + Carboplatin/Paclitaxel: Sym004 administered as an intravenous infusion at a dose 6 mg/kg weekly until unacceptable toxicity, progressive disease, withdrawal of consent, or until the subject met any of the criteria for subject withdrawal, or withdrawal from the IMP in combination with platinum-doublet chemotherapy regimen of carboplatin/paclitaxel (carboplatin area under the concentration-time curve (AUC) = 6 milligram per millilitre per minute [mg/mL/min] plus paclitaxel 225 mg/m^2 on Day 1 of 3-Week cycle intravenously for a maximum of 6 treatment cycles).
- Part 1: Sym004 6/12 mg/kg + Carboplatin/Paclitaxel: Sym004 administered as an intravenous infusion at a dose 6 mg/kg on Day 1 and 12 mg/kg on Day 8 of a 3-Week cycle until unacceptable toxicity, progressive disease, withdrawal of consent, or until the subject met any of the criteria for subject withdrawal, or withdrawal from the IMP in combination with platinum-doublet chemotherapy regimen of carboplatin/paclitaxel (carboplatin AUC = 6 mg/mL/min plus paclitaxel 225 mg/m^2 on Day 1 of every 3-Week cycle intravenously for a maximum of 6 treatment cycles).
Period: Overall Study
Arm/Group | Part 1: Sym004 6 mg/kg + Cisplatin/Gemcitabine | Part 1: Sym004 6 mg/kg + Cisplatin/Pemetrexed | Part 1: Sym004 6 mg/kg + Carboplatin/Paclitaxel | Part 1: Sym004 6/12 mg/kg + Carboplatin/Paclitaxel
Started | 3 | 6 | 3 | 3
Completed | 3 | 6 | 3 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all 15 subjects who were administered any dose of the trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Sym004 6 mg/kg + Cisplatin/Gemcitabine | Part 1: Sym004 6 mg/kg + Cisplatin/Pemetrexed | Part 1: Sym004 6 mg/kg + Carboplatin/Paclitaxel | Part 1: Sym004 6/12 mg/kg + Carboplatin/Paclitaxel | Total
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (7.05) | 59.1 (6.44) | 58.9 (11.09) | 44.8 (10.86) | 56.7 (9.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 1 | 0 | 3
  Male | 3 | 4 | 2 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Dose Limiting Toxicities (DLTs)
Description: DLT: any National Cancer Institute Common Toxicity Criteria for Adverse Events Version 4.03 Grade 4 hematologic or Grade 3/4 non-hematologic toxicities that occurred during DLT observation period and were considered by Investigator to be at least possibly related to trial treatment, and were confirmed by Safety Monitoring Committee (SMC), with exception of Grade 4 neutropenia for not >5 days; Grade 4 lymphocytopenia/ thrombocytopenia for not >5 days; fatigue/headache lasting < 7 days; nausea/vomiting/diarrhoea lasting not >3 days; asymptomatic Grade 3 increase in liver function tests that resolve to baseline within 7 days; Mucositis >= Grade 3 lasting < 7 days; Grade 3 hyperglycemia that resolves in < 7 days; any laboratory values >Grade 3 without any clinical correlate (resolve within 5 days); Grade 3 skin toxicities that resolve to Grade 2 within 7 days; Grade 3/4 hypomagnesemia that resolves within 5 days. Subjects with DLTs presented based on investigator and SMC decision.
Time Frame: Day 1 to Day 21 of Cycle 1
Population: The dose limiting toxicity set included all 15 subjects in the safety analysis set (SAF) who received all planned trial medication doses during the first 21 days following the first dose of Sym004.
Measure: Number; unit: Subjects
Arm/Group | Part 1: Sym004 6 mg/kg + Cisplatin/Gemcitabine | Part 1: Sym004 6 mg/kg + Cisplatin/Pemetrexed | Part 1: Sym004 6 mg/kg + Carboplatin/Paclitaxel | Part 1: Sym004 6/12 mg/kg + Carboplatin/Paclitaxel
Number analyzed (Participants) | 3 | 6 | 3 | 3
Subjects
  Investigator | 2 | 1 | 1 | 0
  SMC | 2 | 1 | 0 | 0

2. Secondary Outcome: Number of Subjects With Treatment-emergent Adverse (TEAEs), Serious TEAEs, TEAEs Leading to Discontinuation and TEAEs Leading to Death
Description: An adverse event (AE) was defined as any untoward medical occurrence in a subject or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. AEs were considered treatment emergent if they started on or after the day of first administration of the first trial treatment given (Sym004 or one of the individual Platinum-Doublet therapies) or if they worsened after receiving first dose of treatment.
Time Frame: Day 1 up to 28 days after last dose of study drug (up to 53 weeks)
Population: The safety analysis set included all 15 subjects who were administered any dose of the trial medication.
Measure: Number; unit: subjects
Arm/Group | Part 1: Sym004 6 mg/kg + Cisplatin/Gemcitabine | Part 1: Sym004 6 mg/kg + Cisplatin/Pemetrexed | Part 1: Sym004 6 mg/kg + Carboplatin/Paclitaxel | Part 1: Sym004 6/12 mg/kg + Carboplatin/Paclitaxel
Number analyzed (Participants) | 3 | 6 | 3 | 3
subjects
  TEAEs | 3 | 6 | 3 | 3
  Serious TEAEs | 3 | 5 | 3 | 3
  TEAE leading to Discontinuation | 1 | 3 | 0 | 2
  TEAEs Leading to Death | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to 28 days after last dose of study drug (up to 53 weeks)
Arm/Group | Part 1: Sym004 6 mg/kg + Cisplatin/Gemcitabine | Part 1: Sym004 6 mg/kg + Cisplatin/Pemetrexed | Part 1: Sym004 6 mg/kg + Carboplatin/Paclitaxel | Part 1: Sym004 6/12 mg/kg + Carboplatin/Paclitaxel
Serious Adverse Events (participants affected / at risk) | 3/3 | 5/6 | 3/3 | 3/3
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Sym004 6 mg/kg + Cisplatin/Gemcitabine (N=3) | Part 1: Sym004 6 mg/kg + Cisplatin/Pemetrexed (N=6) | Part 1: Sym004 6 mg/kg + Carboplatin/Paclitaxel (N=3) | Part 1: Sym004 6/12 mg/kg + Carboplatin/Paclitaxel (N=3)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0
Device related sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 1
Urinary bladder polyp (Renal and urinary disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Sym004 6 mg/kg + Cisplatin/Gemcitabine (N=3) | Part 1: Sym004 6 mg/kg + Cisplatin/Pemetrexed (N=6) | Part 1: Sym004 6 mg/kg + Carboplatin/Paclitaxel (N=3) | Part 1: Sym004 6/12 mg/kg + Carboplatin/Paclitaxel (N=3)
Anaemia (Blood and lymphatic system disorders) | 3 | 6 | 2 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 1 | 1
Hearing impaired (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 1 | 2
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 3 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Lip oedema (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 5 | 2 | 2
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 3 | 2 | 1
Tongue discolouration (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2 | 1
Asthenia (General disorders) | 1 | 3 | 2 | 1
Chills (General disorders) | 1 | 2 | 0 | 0
Hyperthermia (General disorders) | 0 | 1 | 0 | 0
Impaired healing (General disorders) | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 2 | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 1 | 0
Oedema peripheral (General disorders) | 0 | 2 | 1 | 0
Pain (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 1
Sense of oppression (General disorders) | 0 | 0 | 1 | 0
Thrombosis in device (General disorders) | 1 | 0 | 0 | 0
Xerosis (General disorders) | 0 | 3 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 3 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 3 | 2 | 0
Fungal infection (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Genital infection fungal (Infections and infestations) | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 2 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 1 | 0 | 0
Paronychia (Infections and infestations) | 0 | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 2 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0
General physical condition abnormal (Investigations) | 0 | 1 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 3 | 2 | 1
Neutrophil count decreased (Investigations) | 3 | 5 | 2 | 2
Platelet count decreased (Investigations) | 1 | 3 | 2 | 2
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 2 | 2 | 1
White blood cell count decreased (Investigations) | 2 | 2 | 3 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2 | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 4 | 3 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Clubbing (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebellar syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 3 | 2 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 1 | 1
Polyneuropathy (Nervous system disorders) | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0
Depressive symptom (Psychiatric disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 1
Cystitis noninfective (Renal and urinary disorders) | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary bladder polyp (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0
Genital erythema (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Bradypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 1 | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The trial was prematurely discontinued and Expansion Cohort (Part 2) was not conducted as Sponsor decided to prematurely discontinue the development of Sym004. This decision was not related to any safety or efficacy findings regarding Sym004.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No